CLINICAL TRIAL: NCT07187336
Title: The Efficacy and Safety of Shoulder Motion Style Acupuncture Treatment (MSAT) on in Patients With Shoulder Pain Caused by Traffic Accidents: A Pragmatic Randomized Controlled Trial
Brief Title: A Pragmatic Randomized Controlled Trial: The Efficacy and Safety of Shoulder MSAT on in Patients With Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2025-09
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Pain
Keywords: motion style acupuncture treatment
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Intervention Model Description: A Pragmatic randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder MSAT Group (Experimental): Participants receive integrative Korean medicine treatment plus Shoulder Motion Style Acupuncture Treatment (MSAT).
  MSAT: Acupuncture needles are inserted into the affected shoulder, and the practitioner guides or assists joint movements while the needles are retained. This aims to enhance pain relief and improve mobility.
  Treatment schedule: Once daily, 3 sessions during hospitalization (days 2-4).
  Additional integrative treatments: Acupuncture, pharmacopuncture, Chuna manual therapy, and herbal medicine, all provided as standard care.
  Interventions: Procedure: Integrative Korean Medicine Only Group
- Integrative Korean Medicine Only Group (Experimental): Participants receive integrative Korean medicine treatment only, without MSAT.
  Acupuncture: 6-10 points selected by the practitioner; 15-20 minutes per session.
  Pharmacopuncture: Injection of herbal extracts into acupuncture points.
  Chuna manual therapy: Manual therapy for 10-15 minutes daily.
  Herbal medicine: Decoction extracts packaged in pouches, taken twice daily after meals.
  Treatment schedule: Daily during hospitalization.
  Interventions: Procedure: Shoulder MSAT Group; Procedure: Integrative Korean Medicine Only Group

INTERVENTIONS:
Procedure: Shoulder MSAT Group — Shoulder Motion Style Acupuncture Treatment (MSAT) involves inserting acupuncture needles into specific points around the shoulder joint, then guiding or assisting the patient's shoulder movements while the needles remain in place. This combined technique is intended to maximize acupuncture effects by stimulating both the needles and the joint motion.
  In this study, MSAT will be performed once daily for three consecutive days (hospital days 2-4), in addition to standard integrative Korean medicine treatment (acupuncture, pharmacopuncture, Chuna manual therapy, and herbal medicine). Each MSAT session lasts about 10-20 minutes.
  This distinguishes the intervention from the comparator arm, which receives integrative Korean medicine treatment only, without MSAT.
  Arms: Integrative Korean Medicine Only Group
Procedure: Integrative Korean Medicine Only Group — Participants in this group receive only standard integrative Korean medicine treatments, without MSAT. Treatments include acupuncture (6-10 points, 15-20 minutes per session), pharmacopuncture (injection of herbal extracts at acupuncture points), Chuna manual therapy (10-15 minutes daily), and herbal medicine (oral decoction extracts taken twice daily).
  This arm serves as the comparator to distinguish the additional effects of MSAT, since both groups receive the same integrative Korean medicine but only the experimental arm includes Shoulder MSAT.

SUMMARY:
This study will test the effectiveness and safety of Motion Style Acupuncture Treatment (MSAT) for shoulder pain caused by traffic accidents. About 98 hospitalized patients with acute shoulder pain after a traffic accident will take part.

Participants will be randomly assigned to one of two groups:

MSAT + integrative Korean medicine group (acupuncture, herbal medicine, pharmacopuncture, Chuna therapy, plus MSAT), or

Integrative Korean medicine only group (acupuncture, herbal medicine, pharmacopuncture, Chuna therapy).

MSAT involves inserting needles into the shoulder area and gently moving the joint to improve pain relief and mobility. All treatments used in this study are standard care in Korean medicine.

The main outcomes are pain reduction, shoulder movement, daily function, quality of life, and patient satisfaction. Safety will also be monitored by recording any side effects such as temporary soreness, bruising, or discomfort.

Treatment will be provided during hospitalization (up to 5 days), and patients will be followed up by phone at 2 weeks and 1 month after enrollment.

The results of this trial will help determine whether adding MSAT to standard integrative Korean medicine treatment provides greater benefit for patients with acute shoulder pain after traffic accidents.

DETAILED DESCRIPTION:
This pragmatic randomized controlled trial is designed to evaluate the efficacy and safety of Motion Style Acupuncture Treatment (MSAT) for acute shoulder pain resulting from traffic accidents. Shoulder injuries after motor vehicle accidents often cause pain, restricted range of motion, and functional limitations. While integrative Korean medicine treatments such as acupuncture, pharmacopuncture, Chuna manual therapy, and herbal medicine are commonly used, there is limited high-quality evidence regarding the additional benefits of MSAT for shoulder conditions.

MSAT is a therapeutic technique in which acupuncture needles are inserted into affected areas while the practitioner guides or assists the patient's shoulder movements. This combined approach aims to enhance the analgesic and functional effects of acupuncture.

In this trial, 98 inpatients with acute shoulder pain following a traffic accident will be randomized equally into two groups. One group will receive integrative Korean medicine plus MSAT, and the other will receive integrative Korean medicine alone. MSAT will be performed once daily for three sessions during hospitalization (days 2-4), while both groups will continue standard integrative treatments.

The study will assess clinical effectiveness through changes in shoulder pain intensity, range of motion, functional status, quality of life, and patient global impression of change. Safety will be evaluated by monitoring adverse events during treatment and follow-up.

By comparing outcomes between the two groups, this study aims to provide evidence on whether MSAT offers additional benefit beyond integrative Korean medicine for patients with acute shoulder pain after traffic accidents. The findings are expected to contribute to establishing clinical guidance for safe and effective use of MSAT in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 19 to 70 years

Hospitalized with shoulder pain within 5 days after a traffic accident

Shoulder pain intensity ≥ 5 on the Numeric Rating Scale (NRS) with observed limitation of movement

Able and willing to provide written informed consent

Exclusion Criteria:

Serious conditions causing shoulder pain (e.g., malignant tumor, infection)

Progressive or severe neurological deficits

Recent shoulder surgery or procedure within 3 weeks

Shoulder pain mainly due to non-shoulder disorders (e.g., fibromyalgia, rheumatoid arthritis, gout)

Contraindications to MSAT (e.g., fracture, dislocation, ligament rupture or instability, severe inflammation)

Chronic diseases interfering with assessment (e.g., cardiovascular disease, renal disease, diabetic neuropathy, dementia, epilepsy)

Current use of steroids, immunosuppressants, psychiatric drugs, or other medications that may affect results

Contraindications to acupuncture (e.g., bleeding disorders, anticoagulant use, severe diabetes, severe cardiovascular disease)

Pregnant or planning pregnancy

Severe psychiatric illness

Participation in another interventional clinical trial

Unable to provide informed consent

Any other condition deemed inappropriate by the investigator

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale, NRS | Baseline (Day 2, before treatment) to Day 5 (end of hospitalization).
  Patient-reported shoulder pain intensity on a 0-10 scale (0 = no pain, 10 = worst pain).

SECONDARY OUTCOMES:
Shoulder Range of Motion (ROM) | Baseline, Day 5, 2 weeks, and 1 month after enrollment.
  Active and passive ROM in six directions (flexion, extension, abduction, adduction, internal rotation, external rotation), measured with a goniometer.
Shoulder Pain and Disability Index (SPADI) | Baseline, Day 5, 2 weeks, and 1 month after enrollment.
  13-item questionnaire assessing pain (5 items) and disability (8 items), each scored 0-10; higher scores indicate greater disability.
Quality of Life (EQ-5D-5L) | Baseline, Day 5, 2 weeks, and 1 month after enrollment.
  Standardized instrument assessing mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Patient Global Impression of Change (PGIC) | Day 5, 2 weeks, and 1 month after enrollment.
  7-point scale of overall improvement reported by the patient.
Adverse Events | During hospitalization, and at 2 weeks and 1 month follow-up.
  Any expected or unexpected adverse reactions (e.g., local pain, bruising, systemic reactions) assessed by patient report and investigator observation.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, phD, Principal Investigator — Jaseng Medical Foundation

IPD SHARING:
Plan to Share IPD: No